CLINICAL TRIAL: NCT06956950
Title: Efficacy of Adding Magnesium Sulfate to Bupivacaine in Ultrasound-guided Transmuscular Quadratus Lumborum Block for Postoperative Analgesia in Patients Underdoing Hip Arthroplasty
Brief Title: Magnesium Sulfate in Addition to Bupivacaine in Ultrasound-guided Transmuscular Quadratus Lumborum Block for Post-Operative Analgesia After Total Hip Arthroplasty
Acronym: Mgso4
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Mohammad Abdelsattar Elbagoury, Lecturer of anesthesia, surgical ICU and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36264PR1128/3/25
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pain Score Reduction
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: ultrasound-guided transmuscular quadratus lumborum block using 25 ml of 0.25% bupivacaine + 5 ml 10% magnesium sulfate
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacaine /MgSo4 (Active Comparator): patients will receive ipsilateral single-shot of ultrasound-guided transmuscular quadratus lumborum block using bupivacaine plus MgSo4 after surgery
  Interventions: Drug: Bupivacaine + Magnesium sulfate
- bupivacaine/saline (Active Comparator): patients will receive ipsilateral single-shot of ultrasound-guided transmuscular quadratus lumborum block using bupivacaine plus saline after surgery
  Interventions: Drug: Bupivacaine + saline

INTERVENTIONS:
Drug: Bupivacaine + Magnesium sulfate — ultrasound-guided transmuscular quadratus lumborum block using 25 ml of 0.25% bupivacaine + 5 ml 10% magnesium sulfate
  Arms: bupivacaine /MgSo4
Drug: Bupivacaine + saline — ultrasound-guided transmuscular quadratus lumborum block using 25 ml of 0.25% bupivacaine + 5 ml normal saline
  Arms: bupivacaine/saline

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy of adding magnesium sulfate to bupivacaine in ultrasound-guided transmuscular quadratus lumborum block for postoperative analgesia in adult patients underdoing hip arthroplasty. The main questions it aims to answer are:

* Does Magnesium sulphate lower Pain score (VAS) postoperatively.
* Does Magnesium sulphate lowerTotal opioid consumption postoperatively. and What side effects do participants have when taking Magnesium sulphate? Researchers will compare Magnesium sulphate to a placebo (a look-alike substance that contains no drug) to see if Magnesium sulphate works to lower pain score.

Participants will:

* Take with have ultrasound-guided transmuscular quadratus lumborum block after surgery using bupivacaine with Magnesium sulphate or with placebo
* Followed up 48 hours postoperatively to monitor pain score or any reported side effect.

DETAILED DESCRIPTION:
The quadratus lumborum block (QLB) is an abdominal wall fascial block plane block described for providing perioperative analgesia for abdominal, hip and lower limb surgeries . Opioid-sparing analgesic treatments for hip arthroplasty such as lumbar plexus and femoral nerve blocks, are effective but they carry a high risk of undesirable lower limb motor or muscle weakness. Fascia iliaca block, on the other hand, does not consistently provide adequate pain relief. Quadratus lumborum (QL) block is a relatively new truncal regional block technique that provides effective pain control after upper and lower abdominal surgeries. ersalis fascia laterally. The anterior QL block was also classified as transmuscular approach (in between QL and PM muscles) in earlier studies . Local anesthetic injected between the QL muscle and anterior layer of the thoracolumbar fascia can potentially spread to the thoracic paravertebral (PVB) space.

Magnesium plays an important role in the physiological function of the human body. A large number of studies have reported the safetyand effectiveness of adding magnesium sulfate in various regional anesthesia techniques . Therefore, this prospective randomized controlled study to compare the analgesic efficacy of combining magnesium sulfate with bupivacaine in QLB.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* American Society of Anesthesiology (ASA) class I-III
* Undergoing hip arthroplasty .

Exclusion Criteria:

* Patient refusal.
* Body mass index (BMI) > 40 Kg/m2.
* Allergy to local anesthetics or magnesium sulphate.
* coexisting coagulopathy.
* Local infection at puncture site.
* Severe renal impairment ( eGFR < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
postopeative pain Score | 48 hours postoperatively
  The degree of pain will be assessed after surgery by Visual Analogue Score (score for the severity of pain in the range 0-10, where 0 = no pain and 10 = severe pain) at 6 , 12 , 24 , 48 hours postoperatively.

SECONDARY OUTCOMES:
Total opioid consumption | 48 hours postoperatively
  total morphine consumption after surgery
Time to first rescue analgsic request | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Mohammad Abdelsattar Elbagoury, MD, Principal Investigator — lecturer of anesthesia and surgical ICU and pain medicine
Locations (1):
- Faculty of medicine, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No